CLINICAL TRIAL: NCT05411471
Title: A Phase IIb, Randomized, Open-labeled Trial to Evaluate the Immunogenicity and Safety of One or Two Doses of Booster Vaccine With the COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain in Adults in Hong Kong
Brief Title: Immunogenicity and Safety Study of Booster Vaccine With the COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech (Hong Kong) Limited (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-2009
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (1 dose Omicron Vaccine arm, mRNA vaccine group) (Experimental): 75 participants who have completed two/three doses of mRNA vaccine (prior to this study) will receive one dose COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain(1200 SOU).
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain
- Arm 2 (2 doses Omicron Vaccine arm, mRNA vaccine group) (Experimental): 75 participants who have completed two/three doses of mRNA vaccine (prior to this study) will receive two doses COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain (0,28 days)(1200 SOU).
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain
- Arm 3 (1 dose Omicron Vaccine arm, CoronaVac® group) (Experimental): 75 participants who have completed two/three doses of CoronaVac®(prior to this study) will receive one dose COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain (1200 SOU).
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain
- Arm 4 (2 doses Omicron Vaccine arm, CoronaVac® group) (Experimental): 75 participants who have completed two/three doses of CoronaVac®(prior to this study) will receive two doses COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain (0,28 days)(1200 SOU).
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain

INTERVENTIONS:
Biological: COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain — The COVID-19 vaccine (Vero cell), Inactivated, Omicron Strain was developed by Sinovac Life Science Ltd.The product is a pre-filled syringe or a vial with an extractable volume of 0.5 mL. The antigen content is 1200 SOU/0.5 mL (6 µg/0.5 mL).
  Other Names: COVID-19 Omicron Vaccine

SUMMARY:
This is a randomized, open-labeled, Phase IIb clinical trial.The purpose of this study is to evaluate the immunogenicity and safety of the booster vaccine of using one or two doses of COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain in Adults above 18 Years Old Who Have Completed Two or Three Doses of mRNA Vaccine or CoronaVac®.

DETAILED DESCRIPTION:
This is a randomized, open-labeled, Phase IIb clinical trial of 300 participants aged 18 years and above, who have completed two or three doses of mRNA vaccine or CoronaVac® in Hong Kong for at least 90 days after the last dose. After enrollment, the participants will be assigned to 2 groups according to their previous vaccination (mRNA vaccine group and CoronaVac® group) and then each group will be randomly assigned to two study arms at a ratio of 1:1 to receive one or two booster doses of COVID-19 Vaccine (Vero Cell), Inactivated, Omicron Strain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above, who have received two or three prior doses of mRNA COVID-19 vaccine (Comirnaty®, made by BioNTech/Pfizer) or CoronaVac®, with the last dose given at least 90 days prior to the day of booster vaccination in the present study;
* Evidence of a deep throat saliva (DTS) PCR negative for SARS-COV-2 within 24 hours before enrollment;
* Female participants who have a negative pregnancy test on the day of the first dose of the booster vaccine in the present study, and are not currently breastfeeding;
* The participants are able to understand and sign the informed consent voluntarily before the first dose of booster vaccine in the present study;
* The participants are willing and able to comply with all schedule visits, sample collection, vaccine plan, and other study procedures;
* The participants must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of confirmed or having evidence showing a current infection of SARS-CoV-2 prior to randomization or vaccination;
* Any prior administration of another investigational coronavirus vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Known allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Serious chronic disease, serious cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, hepatorenal disease, malignant tumor, etc.;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Receipt of blood/plasma products or immunoglobulins in the past three months before first vaccination in this study;
* Participation in other studies involving study intervention within 30 days prior to first vaccination in this study;
* Receipt of attenuated live vaccines in the past fourteen days prior to each vaccination in this study;
* Receipt of inactivated or subunit vaccines in the past seven days prior to each vaccination in this study;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc.);
* Acute febrile illness with oral temperature >37.5°C on the day of each vaccination;
* According to the investigator's judgment, the participant has any other factors that might interfere with the results of the clinical trial or pose additional risk to the participant due to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Geometric mean of neutralization antibody titre (GMT) | Day 14 after the last booster dose
  Geometric mean of neutralization antibody titre (GMT) on Day 14 after the last booster dose against the Omicron variant in different groups
Occurrence, intensity, duration, and relationship of solicited local and systemic AEs | 28 days post booster vaccination
  Occurrence, intensity, duration, and relationship of solicited local and systemic AEs for 7 days following each booster dose vaccination and of unsolicited AEs for 28 days post booster vaccination

SECONDARY OUTCOMES:
Seroconversion rate of neutralization antibody | Day 14 after the last booster dose
  Seroconversion rate of neutralization antibody against the omicron variant on Day 14 after the last booster dose in different groups
Seropositivity rate of neutralization antibody | Day 14 after the last booster dose
  Seropositivity rate of neutralization antibody against the omicron variant on Day 14 after the last booster dose in different groups
Occurrence and relationship of SAEs | within 6 months post booster vaccination
  Occurrence and relationship of SAEs within 6 months post booster vaccination.

OTHER OUTCOMES:
Seropositive rate of neutralizing antibody | At 90 days and 183 days after one or two doses of booster vaccination
  Seropositive rate of neutralizing antibody to SARS-CoV-2 at 90 days and 183 days after one or two doses of booster vaccination in different groups
GMT of neutralizing antibody | At 90 days and 183 days after one or two doses of booster vaccination
  GMT of neutralizing antibody to SARS-CoV-2 at 90 days and 183 days after one or two doses of booster vaccination in different groups

CONTACTS AND LOCATIONS:
Overall Officials: Ivan HUNG Fan Ngai, Doctor, Principal Investigator — Gleneagles Hospital HongKong
Locations (1):
- Gleneagles Hospital HongKong, Hong Kong, China